CLINICAL TRIAL: NCT05544461
Title: Piloting a Web-based Personalised Nutrition App (eNutri) with UK University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 41/2022
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Diet Habit; Diet, Healthy; Diet Modification
Keywords: Food frequency questionnaire; Nutrition; Dietary intake; Diet quality; Personalised nutrition
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Masking Description: Due to the nature of the study, the participants and researchers will be unblinded. Although the participants will not be explicitly told which group they are in, they will become aware of their group after completing the eNutri FFQ at baseline. Those randomised to the intervention group will receive their eNutri PN advice and those randomised to the control group will not receive any PN advice from eNutri and therefore know which group they have been allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Those in the intervention group will receive eNutri PN advice after completing the eNutri FFQ at baseline only. At weeks 1 and 3 of the study, participants will also receive coaching emails which includes reminders of their PN advice, questions asking them to reflect on their goal progress (if any), and tips and recipes to help them follow the PN advice.
  Interventions: Behavioral: eNutri personalised nutrition advice
- Control group (No Intervention): Those in the control group will not receive any PN advice from eNutri and hence, will not receive any coaching emails. They will only record their diet using the eNutri FFQ.

INTERVENTIONS:
Behavioral: eNutri personalised nutrition advice — eNutri is a web-based app that administers an FFQ and delivers PN advice to the user. The advice is generated from their responses in the FFQ and considers their sex and dietary restrictions (such as whether they eat meat) so the reports are unique to each participant. This report (referred to as a 'healthy eating report') will also include an interactive component, allowing the participant to reflect on the advice received and set personal healthy eating goals to motivate behaviour change. The messages presented in the report have been developed by the eNutri Team, including a registered dietitian and registered nutritionist and are in line with UK dietary guidelines (primarily the EatWell Guide).
  Arms: Intervention group

SUMMARY:
University students account for 50% of the UK young adult population and dietary assessment of this population is crucial in understanding the dietary changes that may occur as they transition to university and adulthood. At this time, many students will leave home for the first time and become responsible for their dietary intake through food shopping and meal preparation. The limited body of evidence in this population group suggests that starting university may be associated with weight gain and the adoption of unhealthful dietary patterns however the extent of these changes may vary based on gender, cooking ability and grocery budget, to name a few. Furthermore, dietary guidance is not typically given to university students although evidence suggests that personalised nutrition advice based on an individual's habitual dietary intake could help to provide the education and support needed for individuals to adopt a healthier diet.

This student pilot study will test whether providing university students with eNutri personalised nutrition advice (intervention group) has a differential impact on diet quality in UK university students compared with those who do not receive any advice (control group) after a 4-week intervention period. 50 university students will use eNutri to record their dietary intake before being randomly allocated to the control or intervention group. After 4 weeks, both groups will repeat the eNutri food and drink questionnaire. Those in the intervention group will also be invited to complete a follow-up questionnaire after a further 8 weeks.

DETAILED DESCRIPTION:
A minimum of 50 participants will be recruited from the University of Reading and University of Hertfordshire and will be asked to complete the eNutri food frequency questionnaire (FFQ) at pre-baseline (week -4) to capture their non-term time diet. 4 weeks later, the participants will be asked to repeat the questionnaire to capture their usual term time diet. At this time point, participants will be randomly allocated by eNutri to either the personalised nutrition (PN) intervention or control group:

* PN intervention group: participants will receive web-based delivery of the eNutri PN advice tailored to their dietary intake, sex and certain dietary restrictions (such as whether they eat meat); PN advice will be unique to each participant.
* Control group: participants will not receive any PN advice from eNutri.

The study will last for 16 weeks with a 4-week intervention period:

* Week -4 (pre-baseline): participants will use eNutri to complete the eNutri FFQ, to provide self-reported anthropometric measurements (height and weight) and to answer questions on behaviour change, physical activity, computer proficiency, and usability of eNutri (via the system usability scale (SUS)).
* Week 0 (baseline): participants will use eNutri to repeat the eNutri FFQ, to provide self-reported anthropometric measurements (height and weight) and demographic information, and to answer questions on behaviour change and physical activity. Those randomised to the PN group will also receive PN advice about their diet via eNutri and will complete a few short questions about which dietary targets they would like to focus on (if any) over the coming weeks to encourage behaviour change.
* Weeks 1 & 3: participants in the PN group only will receive interactive coaching emails to set new dietary goals, be reminded of their PN advice and receive tips and recipes to help them follow the advice.
* Week 4 (end of study): participants in both groups will use eNutri to repeat the eNutri FFQ, provide self-reported weight, answer questions on physical activity and behaviour change, and provide feedback on the dietary advice received from eNutri (intervention group only).
* Week 12 follow-up: participants in the intervention group will complete a short online questionnaire about the longer-term effects of the eNutri dietary advice received during the study.

ELIGIBILITY:
Inclusion Criteria:

* Solely responsible for their own meal preparation and/or food purchases (includes catered and non-catered students)
* Studying at the University of Reading or University of Hertfordshire, UK
* Student in any year of study
* 18 years or older
* Able to read and understand written English without difficulties
* Able to access eNutri using a suitable device (laptop, computer, tablet, or smartphone) with access to the internet
* Have an active email address
* Willing to complete online questionnaires and interact with eNutri on multiple occasions

Exclusion Criteria:

* Students who are not studying full time in-person at university in the academic year 2022-2023 (e.g., part-time students, apprenticeship students or those on a work placement)
* Students whose food choices are in part influenced/determined by others (e.g., students who live with parents, partner, or children during term time, including those who return home every weekend)
* Those reliant on meals where there is limited choice/alternative options (e.g., Recipe boxes such as Gousto, Hello Fresh and Mindful Chef, or those who eat frozen meals brought from home); catered students can take part.
* Pregnant, lactating or planning a pregnancy within the next 4 months
* Food allergies to dairy, nuts/seeds and/or fish/shellfish
* Medical conditions/treatments that have a considerable impact on an individual's diet/appetite on a day-to-day basis (e.g., severe gastrointestinal disorders)
* Have a current or previously diagnosed eating disorder
* Usually eat on fewer than 2 occasions per day
* Receiving dietary advice from a dietitian, nutritionist or medical professional or plan to do so within the next 4 months
* Following a restrictive diet, such as a vegan diet, sport's nutrition diet, meal replacement shake/juice diet (e.g., SlimFast), intermittent fasting diet (e.g,. 5:2), very low carbohydrate diet (e.g., keto, Atkins) or any "fad"/"celebrity" diet, or plan to do so within the next 4 months; vegetarians can take part.
* Following a weight-loss programme, such as Weight Watchers, Noom, LighterLife and Slimming World, or plan to do so within the next 3 months; those aiming to lose weight through general healthy eating and "cutting down" without following specialised weight loss advice can take part.
* Taking weight-loss medication (prescribed or over the counter) or plan to do so within the next 3 months.
* Visual and/or physical impairments that prevent an individual from interacting with visual elements on the screen on their device/using their device, such as clicking buttons/mouse or using the touch pad or viewing images.
* Taking part in another nutrition-related research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Diet quality score (DQS) | Baseline
  An 11-item eNutri DQS will be automatically calculated by eNutri after completing the FFQ. The eNutri DQS was developed for Northern European adults and quantifies diet quality (i.e. the healthiness of a diet). It is composed of 11 food and nutrient components that are summed to give an overall score, where higher scores reflect the healthiest diets based on adherence to dietary guidelines
Diet quality score (DQS) | Week 4
  An 11-item eNutri DQS will be automatically calculated by eNutri after completing the FFQ. The eNutri DQS was developed for Northern European adults and quantifies diet quality (i.e. the healthiness of a diet). It is composed of 11 food and nutrient components that are summed to give an overall score, where higher scores reflect the healthiest diets based on adherence to dietary guidelines

SECONDARY OUTCOMES:
Weight | Pre-baseline
  Self-reported measurement of weight
Weight | Baseline
  Self-reported measurement of weight
Weight | Week 4
  Self-reported measurement of weight
Height | Pre-baseline
  Self-reported measurement of height
Height | Baseline
  Self-reported measurement of height
Body mass index (BMI) | Pre-baseline
  Automatically calculated by eNutri after providing self-reported weight and height
Body mass index (BMI) | Baseline
  Automatically calculated by eNutri after providing self-reported weight and height
Body mass index (BMI) | Week 4
  Automatically calculated by eNutri after providing self-reported weight and height
eNutri Food Frequency Questionnaire (FFQ) dietary intake data | Pre-baseline (week -4)
  eNutri includes a 157-item FFQ which participants will use to identify how often they typically ate/drank each item during the last 4 weeks (e.g. once a day, less than once a week, not in the last 4 weeks) then choose their typical portion size from a range of 7 photos/buttons. To increase the accuracy of the FFQ, some food/drink items have an extra question, such as the type of milk used on breakfast cereals/hot drinks or whether the food/drink item consumed was a reduced fat/sugar variety. The responses to the FFQ are used to automatically calculate the average intake in grams per day for each food item.
eNutri Food Frequency Questionnaire (FFQ) dietary intake data | Baseline
  eNutri includes a 157-item FFQ which participants will use to identify how often they typically ate/drank each item during the last 4 weeks (e.g. once a day, less than once a week, not in the last 4 weeks) then choose their typical portion size from a range of 7 photos/buttons. To increase the accuracy of the FFQ, some food/drink items have an extra question, such as the type of milk used on breakfast cereals/hot drinks or whether the food/drink item consumed was a reduced fat/sugar variety. The responses to the FFQ are used to automatically calculate the average intake in grams per day for each food item.
eNutri Food Frequency Questionnaire (FFQ) dietary intake data | Week 4
  eNutri includes a 157-item FFQ which participants will use to identify how often they typically ate/drank each item during the last 4 weeks (e.g. once a day, less than once a week, not in the last 4 weeks) then choose their typical portion size from a range of 7 photos/buttons. To increase the accuracy of the FFQ, some food/drink items have an extra question, such as the type of milk used on breakfast cereals/hot drinks or whether the food/drink item consumed was a reduced fat/sugar variety. The responses to the FFQ are used to automatically calculate the average intake in grams per day for each food item.
Individual DQS component scores, food group intakes (e.g. vegetables, wholegrains) and nutrient intakes (e.g. saturated fat, sodium) | Pre-baseline (Week -4)
  Recorded via eNutri FFQ
Individual DQS component scores, food group intakes (e.g. vegetables, wholegrains) and nutrient intakes (e.g. saturated fat, sodium) | Baseline
  Recorded via eNutri FFQ
Individual DQS component scores, food group intakes (e.g. vegetables, wholegrains) and nutrient intakes (e.g. saturated fat, sodium) | Week 4
  Recorded via eNutri FFQ
Usability of eNutri measured by the System Usability Scale (SUS) | Baseline
  The SUS is a 10-item questionnaire with 5 response options that range from Strongly Agree to Strongly Disagree and is a reliable tool for measuring usability.
Participants motivation and perceived ability to make dietary changes | Pre-baseline (Week -4)
  Measured through a short psychology questionnaire covering ability, opportunity, motivation, and knowledge
Participants motivation and perceived ability to make dietary changes | Baseline
  Measured through a short psychology questionnaire covering ability, opportunity, motivation, and knowledge
Participants motivation and perceived ability to make dietary changes | Week 4
  Measured through a short psychology questionnaire covering ability, opportunity, motivation, and knowledge
Participant feedback on the dietary advice received from eNutri | Week 4
  Questionnaire covering how effective the dietary advice was at encouraging the participants to make healthy changes to their diet and whether they encountered any barriers (intervention group only).
Feedback on the longer-term impact of the dietary advice received from eNutri | Week 12
  A follow-up questionnaire provided at week 12 to determine whether there was a longer-term impact of the dietary advice received (intervention group only).

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lovegrove, Professor, Principal Investigator — Hugh Sinclair Unit of Human Nutrition, University of Reading
Locations (2):
- United Kingdom (2):
  - University of Reading, Reading, Berkshire
  - University of Hertfordshire, Hatfield, Hertfordshire

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymised individual participant data that underlie results in publications in a public repository. Sharing of IPD will be in line with the confidentiality and consent agreements. This may include:
  * Sociodemographics
  * Anthropometrics
  * Dietary intake data
Time Frame: No later than the time of first publication and available indefinitely thereafter.
Access Criteria: We plan for open access.

REFERENCES:
- [Background] Zenun Franco R, Fallaize R, Weech M, Hwang F, Lovegrove JA. Effectiveness of Web-Based Personalized Nutrition Advice for Adults Using the eNutri Web App: Evidence From the EatWellUK Randomized Controlled Trial. J Med Internet Res. 2022 Apr 25;24(4):e29088. doi: 10.2196/29088. PMID 35468093